CLINICAL TRIAL: NCT05305144
Title: Identification and Evaluation of Micro-vascular Retinal and Brain Markers to Establish Potential Early Brain Structural Alterations in Young Adults - SHIVA-Share
Brief Title: Retinal, Cerebral and Vascular Precursor Markers of Cerebral Small Vessel Disease.
Acronym: SHIVA-SHARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: University of Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2020/42
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: Cognitive decline; dementia; stroke; small vessel disease; brain imaging; adaptive optics; optical coherence tomography angiography; prevention; risk prediction
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Cognitive Dysfunction; Dementia; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ophthalmological and vascular assessments (Experimental): This single-center national interventional study aims to collect ophthalmological (retinal image acquisition) and blood pressure (vascular assessment) data from 400 young adults from the Bordeaux bio-Share cohort, during two visits taking place one year apart.
  Interventions: Procedure: Vascular and ophthalmological examinations

INTERVENTIONS:
Procedure: Vascular and ophthalmological examinations — Part. 1 - Vascular checkup examinations:
  After collecting classic clinical parameters (weight, height, waist circumference), the in-depth vascular workup of each participant will include the following measurements:
  * Measurement of central arterial pressure,
  * Measurement of arterial stiffness,
  * Continuous blood pressure measurement (beat-to-beat),
  * Heart rate measurement,
  * 24-hour blood pressure measurement with QKD (holter).
  Part. 2 - Ophthalmological examinations:
  After dilating the pupil, a series of examinations will be conducted on the participant:
  * Auto-refractometry
  * Measurement of the axial length of the globe
  * Color retinophotography of the retina,
  * Adaptive Optics Exam
  * SS-OCT-A exam

SUMMARY:
Cognitive impairment and dementia are primarily due to a combination of vascular brain injury and neurodegenerative lesions. The vascular component is now recognized as a major contributor to the pathophysiology of dementia, with small vessel disease (SVD) being its most frequent substrate. This study aims to collect retinal microvascular markers as well as various parameters related to blood pressure and arterial stiffness, in a young adult population. The main objective is to explore the association between these parameters and structural changes on brain MRI. Results will allow to determine the most relevant biomarkers associated with very early brain imaging markers of SVD.

DETAILED DESCRIPTION:
Small Vessel Disease is most often covert i.e detectable only on brain images without being associated with a clinical stroke. Covert SVD (cSVD) is highly prevalent in older persons from the general population and is a powerful predictor of future cognitive decline and dementia risk. Better detection of covert cSVD, particularly at the earliest stages, would have a major impact on preventing disability and costs related to stroke, cognitive impairment and dementia. Studying the association of retinal and vascular biomarkers with MRI markers of brain structure will enable to facilitate the detection of patients at high risk of developing cSVD and its complications. This study aims to collect ophthalmological (retinal image acquisition - Part 1 of the study) and blood pressure / arterial stiffness (vascular assessment - Part 2 of the study) markers from 400 young adults from the Bordeaux bio-Share study. In Part 1, microvascular retinal biomarkers will be revealed by two complementary advanced technologies: the Swept-source optical coherence tomography angiography (SS-OCT-A) and the Adaptative Optics (AO). In Part 2, participants will benefit from an in-depth vascular assessment.

ELIGIBILITY:
Inclusion Criteria: Young adults from the i-Share cohort will be included in the study:

* having signed the informed consent form of the MRi-Share sub-study,
* having signed the informed consent form for the bio-Share sub-study,
* for whom brain MRI images and for whom the results of the genome-wide genetic association study (GWAS) are of good quality
* having signed freely, an informed and written consent for this study (at the latest on the day of inclusion and before any examination required by the research),
* being affiliated with social security.

Exclusion Criteria: Will not be included in the study:

* participants with severe myopia greater than -6 dioptres
* participants with known allergy to Tropicamide (Mydriaticum®)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2024-06-07 (Estimated); Study Completion 2024-06-07 (Estimated)

PRIMARY OUTCOMES:
Part 1 VASCULAR PARAMETERS RELATED TO BLOOD PRESSURE - Central arterial pressure by carotid tonometry (systolic, diastolic, mean) | within the inclusion visit (at the time of the vascular assessment)
  Central arterial pressure by carotid tonometry (systolic, diastolic, mean)

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie DEBETTE, Pr, Principal Investigator — INSERM U1219 Bordeaux Population Health
Locations (1):
- CHU de Bordeaux, Bordeaux, France